CLINICAL TRIAL: NCT02673567
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Pharmacokinetics, Safety, and Tolerability of Single Doses Subcutaneous Administration of TEV-48125 (Doses up to 900 mg) in Japanese and Caucasian Healthy Subjects
Brief Title: To Assess Pharmacokinetics, Safety and Tolerability of TEV-48125 in Japanese and Caucasian Healthy Subjects After a Single Subcutaneous (SC) Administration of TEV-48125
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TV48125-PK-10078
Record Dates: First submitted 2016-01-26; First posted 2016-02-04 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Antibodies, Monoclonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TEV-48125 - 1 (Experimental): Dose Regimen 1
  Interventions: Drug: TEV-48125 - 1
- TEV-48125 - 2 (Experimental): Dose Regimen 2
  Interventions: Drug: TEV-48125 - 2
- TEV-48125 - 3 (Experimental): Dose Regimen 3
  Interventions: Drug: TEV-48125 - 3
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-48125 - 1 — Subcutaneous administration Dose Regimen 1
  Other Names: monoclonal antibody
  Arms: TEV-48125 - 1
Drug: TEV-48125 - 2 — Subcutaneous administration Dose Regimen 2
  Other Names: monoclonal antibody
  Arms: TEV-48125 - 2
Drug: TEV-48125 - 3 — Subcutaneous administration Dose Regimen 3
  Other Names: monoclonal antibody
  Arms: TEV-48125 - 3
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled study to assess the pharmacokinetics, safety, and tolerability of subcutaneous administration of TEV-48125 (single ascending doses and single doses up to 900 mg) in Japanese and Caucasian healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a man or woman, 18 to 55 years of age, inclusive
* The subject has a body mass index (BMI) ranging from 17.5 to 28.0 kg/m2, inclusive
* The subjects must be in a good health at screening and check-in

Additional inclusion criteria for Japanese subjects:

* Subject must be a non-naturalized Japanese citizen and hold a Japanese passport
* Subject must have/had 2 Japanese parents and 4 Japanese grandparents who are all non naturalized Japanese citizens
* Subject has been living outside of Japan for no more than 10 years

Additional inclusion criteria for Caucasian subjects:

* The subject has/had 2 Caucasian parents and 4 Caucasian grandparents. Caucasian includes White and Hispanic ethnicities.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The subject is a woman who is pregnant or lactating
* The subject is suffering from, or has a clinically significant history of, 1 or more of the following: cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, hematologic or psychiatric disorder(s)
* The subject has a known allergy or sensitivity to injected proteins, including monoclonal antibodies, or any other component of the formulation. In addition, presence of history of allergies requiring acute or chronic treatment
* Precipitation in another clinical study of a new investigational drug within 30 days (90 days for biologics) before dosing

  * Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | 33 weeks
Time to maximum observed plasma drug concentration (tmax) | 33 weeks
AUC from time 0 to the time of the last measurable plasma drug concentration (AUC0-t) | 33 weeks
AUC from time 0 to 672 hours (4 weeks) postdose (AUC0-672) | 33 weeks
AUC from time 0 extrapolated to infinity (AUC0-∞) | 33 weeks
Percentage extrapolated AUC (%AUCext) | 33 weeks
Apparent serum terminal elimination rate constant (λz) | 33 weeks
Apparent total body clearance (CL/F) | 33 weeks
Apparent volume of distribution during the terminal phase (Vz/F) | 33 weeks
Apparent serum terminal elimination half-life (t½) | 33 weeks

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | 33 weeks
Tolerability- Percentage of participants who fail to complete the study | 33 weeks
Percentage of participants who fail to complete the study due to adverse events | 33 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 13529, Glendale, California, United States